CLINICAL TRIAL: NCT05745389
Title: CorEvitas Alopecia Areata (AA) Safety and Effectiveness Registry
Status: Recruiting | Type: Observational
Sponsor: CorEvitas (Network)
Responsible Party: Sponsor
Other Study IDs: CorEvitas-AA-560
Record Dates: First submitted 2023-02-16; First posted 2023-02-27 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-01

CONDITIONS: Alopecia Areata
MeSH Terms: conditions — Alopecia Areata

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Alopecia Areata: Pts presenting to enrolling sites across the US are invited to enroll if eligible

SUMMARY:
Prospective, observational cohort study for subjects with AA under the care of a dermatology provider. Approximately 5,000 subjects and 100 clinical sites in North America will be recruited to participate with no defined upper limit for either target.

DETAILED DESCRIPTION:
The objective of the registry is to create a cohort of AA subjects to study long-term safety and effectiveness of AA treatments. Because the long-term understanding of safety and efficacy is still limited even after regulatory approval,enrollment and long-term follow-up of a large number of diverse real-world patients exposed to therapies of interest is important to understand safety and effectiveness. The observational structured data collected will be used to better characterize the natural history of the disease and to extensively evaluate the effectiveness and safety of medications approved for the treatment of AA to support ongoing risk benefit evaluation by drug manufacturers and regulators.Further, data collected will inform clinical decision making by subjects and treating providers. This will be done through the standardized collection of validated patient-reported outcomes (PRO) and clinician-reported outcomes (ClinRO), the active evaluation of prevalent and incident comorbidities and adverse events, and the recording of medication utilization patterns. Personal information is also collected from each consenting registry subject allowing for linkages to other public or private clinical and administrative databases, as well as to databases maintained by organizations focused on the care and treatment of AA for the purposes of clinical, market, or outcomes research. This provides an opportunity to evaluate other aspects of the disease and its treatment including but not limited to clinical and drug cost-effectiveness, health care resource utilization, and subject adherence.

ELIGIBILITY:
Inclusion Criteria:

* A subject must meet all the following criteria to participate in the registry:

  1. Has been diagnosed with alopecia areata by a dermatologist or a qualified dermatology practitioner.
  2. Is at least 18 years of age or older.
  3. Is willing to provide Personal Information.
  4. Is prescribed or starting an Enrollment Eligible Medication at the time of enrollment.

Exclusion Criteria:

* Any of the following would exclude the subject from participating in the registry:

  1. Is participating or planning to participate in a double-blind randomized trial for an AA drug. Note:

Concurrent participation in another observational registry or open-label Phase 3b/4 trial is allowed.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients are enrolled in the AA Registry during regularly scheduled office visits. Selected dermatologists are invited to participate as investigators in the Registry.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2022-10-25 (Actual); Primary Completion 2099-12-31 (Estimated); Study Completion 2099-12-31 (Estimated)

PRIMARY OUTCOMES:
Alopecia epidemiology, presentation, natural history, management, and outcomes | A minimum of 10 years from last patient enrolled
  The major clinical outcomes include an assessment of the epidemiology of AA; to better understand the presentation, natural history, management and outcomes.

SECONDARY OUTCOMES:
Physician Reported - Skindex-16 | every 6 months for 10 years
Physician Reported - Alopecia Areata Symptom Impact Scale (AASIS) | every 6 months for 10 years
Physician Reported - Dermatology Life Quality Index (DLQI) | every 6 months for 10 years
Physician Reported - Severity of Alopecia Tool (SALT) | every 6 months for 10 years
Physician Reported - Alopecia Areata-Investigator Global Assessment (AA-IGA) | every 6 months for 10 years
Physician Reported - ClinRo Measure for Eyebrow, Eyelash Hair Loss & Nail Appearance | every 6 months for 10 years
Physician Reported - Alopecia Areata Scale (AAS) | every 6 months for 10 years
Patient Reported - Scalp Hair Assessment PRO | every 6 months for 10 years
Patient Reported - PRO Measure for Eyebrows, Eyelashes & Nail Apperance | every 6 months for 10 years
Patient Reported - Work Productivity and Activity Impairment (WPAI) | every 6 months for 10 years

CONTACTS AND LOCATIONS:
Locations (1):
- CorEvitas, LLC, Waltham, Massachusetts, United States